CLINICAL TRIAL: NCT06560398
Title: Working Through Outreach, Navigation and Digital Enabled Referral and Recruitment Strategies (ACT WONDER²S)
Acronym: ACT WONDER²S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCC-22140; U01CA274971-01 (NIH)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Catchment Area Priority Zone (CAPZ) Intervention - Community Residents and Moffitt Patients (Experimental): Study interventions will be deployed in geographically defined intervention priority zones including Clinical Trial Education sessions and the ACT WONDER²S Phone-line/Email. Community residents in these zones may be exposed to these interventions.
  Residents who are also new patients to Moffitt may be exposed to the CHOICES DA website once they are registered at Moffitt.
  Interventions: Behavioral: Clinical Trial Education Sessions (Community Residents Only); Behavioral: ACT WONDER²S Phone-line/Email (Community Residents and Moffitt Patients); Behavioral: New Patient Information (Moffitt Patients Only)
- Catchment Area Priority Zone (CAPZ) Control - Community Residents and Moffitt Patients (Active Comparator): Study interventions will not be deployed in the control priority zones. Community residents in these zones are unlikely to be exposed to any of the study interventions.
  Interventions: Other: No Intervention
- Catchment Area Priority Zone (CAPZ) Intervention - Community Physicians (Experimental): Study interventions will be deployed in geographically defined intervention priority zones including Continuing Medical Education events, the Trial Connect Portal, and Clinical Trial Newsletters. Community physicians in these zones may be exposed to these interventions.
  Interventions: Behavioral: Continuing Medical Education Events (CME); Behavioral: Trial Connect Portal; Behavioral: Clinical Trial Newsletters
- Catchment Area Priority Zone (CAPZ) Control- Community Physicians (Active Comparator): Study interventions will not be deployed in the control priority zones. Community physicians in these zones are unlikely to be exposed to any of the study interventions.
  Interventions: Other: No Intervention
- Cancer Center Clinical Research Coordinators (CRCs) (Experimental): CRCs that work on therapeutic clinical trials at Moffitt will have access to the implicit bias educational module and digital tools to monitor and enhance minority recruitment, including the Trial Connect Portal and Recruitment Dashboard.
  Interventions: Behavioral: Trial Connect Portal; Behavioral: Implicit Bias Training; Behavioral: Recruitment Dashboard
- Cancer Center Physicians (Experimental): Physicians at Moffitt will have access to the implicit bias educational module and to digital tools to monitor and enhance minority recruitment, including the Trial Connect Portal, Recruitment Dashboard, Portfolio Profiler, and the Eligibility Criteria Calculator.
  Interventions: Behavioral: Trial Connect Portal; Behavioral: Implicit Bias Training; Behavioral: Recruitment Dashboard; Behavioral: Portfolio Profiler; Behavioral: Eligibility Calculator

INTERVENTIONS:
Behavioral: Continuing Medical Education Events (CME) — An engaging 1-hour informational session focusing on topic areas such as implicit bias and emerging evidence from recent cancer clinical trials with CME credit or American Board of Internal Medicine (ABIM) Maintenance of Certification (MOC) points available.
  Arms: Catchment Area Priority Zone (CAPZ) Intervention - Community Physicians
Behavioral: Trial Connect Portal — A digital tool to help facilitate rapid referral of patients to clinical trial opportunities at Moffitt.
  Arms: Cancer Center Clinical Research Coordinators (CRCs); Cancer Center Physicians; Catchment Area Priority Zone (CAPZ) Intervention - Community Physicians
Behavioral: Clinical Trial Newsletters — Electronic/paper newsletters to highlight open trials at Moffitt that will be distributed by email/mail.
  Arms: Catchment Area Priority Zone (CAPZ) Intervention - Community Physicians
Behavioral: Implicit Bias Training — A one-hour educational module will cover information on implicit bias to support the recruitment of diverse patients.
  Arms: Cancer Center Clinical Research Coordinators (CRCs); Cancer Center Physicians
Behavioral: Recruitment Dashboard — A dynamic dashboard depicting the number of patients recruited to clinical trials by gender, race, ethnicity, age, cancer type, residence in the catchment area, and other key clinical characteristics.
  Arms: Cancer Center Clinical Research Coordinators (CRCs); Cancer Center Physicians
Behavioral: Portfolio Profiler — An interactive dashboard to allow cancer center physicians easily identify gaps in the current clinical trial portfolio that may be contributing to racial/ethnic disparities in trial enrollment.
  Arms: Cancer Center Physicians
Behavioral: Eligibility Calculator — A digital calculator that will allow for assessment of the potential impact of clinical trial eligibility criteria (e.g., comorbidities, age, lab values) that may disproportionately exclude patients who are Black and Hispanic prior to submission of clinical trial protocols to the Scientific Review Committee.
  Arms: Cancer Center Physicians
Behavioral: Clinical Trial Education Sessions (Community Residents Only) — An engaging 1-hour educational session delivered by a community health educator that includes basic information about clinical trials, their importance, myths, need for diversity in the trials process, and resources for finding more information about clinical trials.
  Arms: Catchment Area Priority Zone (CAPZ) Intervention - Community Residents and Moffitt Patients
Behavioral: ACT WONDER²S Phone-line/Email (Community Residents and Moffitt Patients) — A study team member will be available for questions via a dedicated phone-line and email for community residents and Moffitt patients with a return contact within 24-hours.
  Arms: Catchment Area Priority Zone (CAPZ) Intervention - Community Residents and Moffitt Patients
Behavioral: New Patient Information (Moffitt Patients Only) — Including CHOICES DA, a web-based tool to improve multiple aspects of decision-making related to participation in cancer clinical trials.
  Arms: Catchment Area Priority Zone (CAPZ) Intervention - Community Residents and Moffitt Patients
Other: No Intervention — Control group with no intervention.
  Arms: Catchment Area Priority Zone (CAPZ) Control - Community Residents and Moffitt Patients; Catchment Area Priority Zone (CAPZ) Control- Community Physicians

SUMMARY:
The purpose of the study is to refine, finalize, implement, and evaluate a multi-level intervention aimed at increasing enrollment of Black and Hispanic patients to National Cancer Institute (NCI)-sponsored therapeutic clinic trials at Moffitt Cancer Center.

DETAILED DESCRIPTION:
A stratified cluster randomized design will be used to assess the impact of the Advancing Clinical Trials: Working through Outreach, Navigation, and Digitally Enabled Referral and Recruitment Strategies (ACT WONDER²S) multi-level intervention on increasing referral and enrollment to NCI-sponsored therapeutic clinical trials among Black and Hispanic patients. Geospatial analytics were used to identify clusters of census tracts within the Moffitt catchment area ("priority zones") with high Black and Hispanic populations for intervention deployment. Priority zones were then matched on population characteristics and randomized to receive the intervention (n=7) or to serve as controls (n=7).

External target populations within the Catchment Area Priority Zone (CAPZ) include community residents and community physicians, while internal target populations within Moffitt Cancer Center (Moffitt) include physicians, clinical research coordinators (CRCs), and patients. The outreach and education intervention components will be facilitated by community health educators (CHEs) targeting community residents (Clinical Trial Education module and CHE support through the ACT WONDER²S Phone-line/Email), community physicians (Continuing Medical Education sessions including implicit bias training), patients at Moffitt (CHE support) and cancer center physicians/CRCs (an implicit bias training). Digitally enabled decision support tools will be developed and deployed to the CHE's (a data-empowered interactive map for outreach planning [Precision Engagement Tool]), community physicians (Clinical Trial Newsletters), patients at Moffitt (a clinical trial decision aid [CHOICES DA]), and cancer center physicians/CRCs (a recruitment dashboard to monitor clinical trial accrual rates, a clinical trial portfolio profiler, and a tool to assess the impact of clinical trial inclusion/exclusion criteria on eligibility across patient populations defined by age, race, and ethnicity [Eligibility Criteria Calculator]). In addition, an online portal (called the Trial Connect Portal) will be developed to connect community-based referring physicians to information about MCC trials and to facilitate their communication with cancer center physicians and CRCs. The primary outcome, enrollment to clinical trials, will be measured by comparing the percentage of Moffitt patients enrolled on NCI-supported treatment trials who are Black or Hispanic between intervention priority zones and the control priority zones. The secondary outcome, referral to Moffitt, will be measured by comparing the percentage of patients referred to Moffitt who are Black or Hispanic between the intervention priority zones and the control priority zones.

ELIGIBILITY:
Inclusion Criteria:

* Community residents: Community residents may engage with various intervention components deployed in the intervention priority zones.
* Community Physicians: may engage with various intervention components deployed in the intervention priority zones if they 1) practice medicine in one of the geographic priority zones.
* Cancer Center Physicians: may engage with various intervention components if they 1) practice medicine at Moffitt.
* Clinical Research Coordinators (CRC): may engage with various intervention components if they 1) work as a CRC at Moffitt and 2) coordinate/pre-screen patients for at least 1 therapeutic clinical trial at Moffitt.
* Cancer Center Patients: may engage with various intervention components if they have an address that maps to an intervention priority zone and 2) are newly registered patients or new existing patients (NEPs).

Exclusion Criteria:

* Community residents, Community Physicians, Cancer Center Physicians, Clinical Research Coordinators, and Moffitt patients who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7649 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment of Black and Hispanic Patients to NCI-sponsored cancer treatment clinical trials | 2 years
  Intervention impact on enrollment rates will be measured by comparing the percentage of Moffitt patients enrolled on NCI-supported treatment trials who are Black or Hispanic between intervention priority zones and the control priority zones.

SECONDARY OUTCOMES:
Referral of Black and Hispanic Patients to Moffitt Cancer Center | 2 Years
  Intervention impact on referral rates will be measured by comparing the percentage of patients referred to Moffitt who are Black or Hispanic between the intervention priority zones and the control priority zones.
Community residents in the intervention CAPZ | 2 years
  The number of community residents that attend a CT educational session.
Community physicians in the intervention CAPZ | 2 years
  The number of physicians that attend a CME event.
Cancer Center CRC | 2 years
  The number of CRCs that used at least one of the CT digital tools.
Cancer Center Physician | 2 years
  The number of MCC physicians that used at least one of the CT digital tools.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Vadaparampil, PhD, Principal Investigator — Moffitt Cancer Center; Dana Rollison, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States